CLINICAL TRIAL: NCT05547906
Title: An Open-label, Dose-escalation, Dose-expansion, Phase 1 Study to Evaluate the Tolerability, Safety, Pharmacokinetics/Pharmacodynamics, and Antitumor Effect of ASCA101 in Patients With Advanced Solid Tumors
Brief Title: Evaluation of the Safety and Efficacy of ASCA101 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MetaFines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MF-ASCA101-01
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ASCA101 IV (Experimental): The study drug, ASCA101(300mg/vial), will be reconstituted in water for injection and diluted with saline to a dose calculated according to individual body surface area or body weight.
  Interventions: Drug: ASCA101

INTERVENTIONS:
Drug: ASCA101 — IV infusion Twice a Week, 8 times per each Cycle

SUMMARY:
This is a prospective, open-label, dose escalation Phase 1 study. The purpose of this study is to evaluate the following objectives in patients with advanced solid tumors after failure of standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years with pathologically or cytologically confirmed metastatic or unresectable advanced solid tumors that progressed despite standard of care or which did not tolerate standard of care and for which other standard of care is not available.
2. Patients with the following laboratory test values, obtained within 14 days prior to study enrollment with no history of G-CSF or blood transfusions within 14 days prior to collection of samples for the laboratory tests:

   * ANC ≥ 1,500/mm³

     * Platelet count ≥ 100,000/mm³

       * Hemoglobin ≥ 9.0 g/dL

         * CrCl ≥ 60 mL/min calculated using the Cockcroft-Gault formula ⑤ Total bilirubin ≤ 1.5×ULN ⑥ AST, ALT ≤ 3×ULN (≤ 5×ULN for patients with liver metastasis or liver cell carcinoma) ⑦ INR and aPTT ≤ 1.5×ULN ⑧ Urine protein to creatinine ratio (UPC) < 1.0 (g/g)a a UPC will be performed in patients with at least one positive (+) protein outcome upon urinalysis.
3. At least one evaluable lesion based on the response evaluation criteria in solid tumors (RECIST) version 1.1 as measured by tumor markers or CT/MRI.
4. Life expectancy ≥ 12 weeks.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Women of childbearing potential who test negative for pregnancy (by serum-hCG or urine-hCG at the discretion of the investigator) at the time of study participation (i.e., all women who have had menarche and are not surgically sterile [hysterectomy, bilateral tubal ligation, bilateral ovariectomy, etc.] and are not post-menopausal [no menstruation for ≥ 12 months for no other medical reasons]).
7. Patients who agree to use medically acceptable methods of birth control (patient's or partner's vasectomy, tubal ligation, intrauterine device, barrier contraception, oral contraceptives, diaphragm or condom use in combination) during treatment with the investigational product (IP) and for 6 months after the end of treatment.
8. Patients who voluntarily provide written informed consent to participate in the study.

Exclusion Criteria:

1. History of hypersensitivities to any of the components of the IP or the same class of drugs as the IP.
2. At the time of the 1st treatment:

   * < 4 weeks from a major surgery, if applicable
   * < 2 weeks from a minor surgery, if applicable
   * < 3 weeks from the last radiotherapy, if applicable
   * < 5 x half-life or < 3 weeks, whichever is longer, from chemotherapy or hormone therapy, if applicable (those who were treated with nitrosoureas or mitomycin within 6 weeks prior to the 1st treatment or targeted biological antibodies within 4 weeks prior to the 1st treatment were not allowed to participate in the study.)
   * < 4 weeks from anticancer immunotherapy, if applicable
3. History of cardiovascular disorders within the past 5 years:

   * New York heart association (NYHA) class ≥ II (or left ventricle ejection fraction ≤ 50%) congestive heart failure (CHF)
   * Uncontrolled hypertension (systolic blood pressure [SBP]/diastolic blood pressure [DBP] > 140/90 mmHg)
   * History of hypertensive crisis or hypertensive encephalopathy
   * Pulmonary hypertension
   * Myocardial infarction
   * Significant vascular disease (e.g., aortic aneurysm requiring surgery or recent peripheral artery thrombosis) within 6 months prior to IP initiation
   * Uncontrolled arrhythmia
   * QTcF interval > 470 msec on screening electrocardiogram (ECG)
4. Clinically significant NCI-CTCAE v5.0 Grade ≥ 1 (allowing Grade ≥ 2 alopecia) ongoing toxicities from previous anticancer treatment.
5. Severe infection or severe traumatic systemic disorders.
6. Symptomatic or uncontrolled metastasis to central nervous system (CNS) (a patient with asymptomatic CNS metastasis may participate in the study if systemic corticosteroids were discontinued ≥ 4 weeks prior and the patient is radiologically and neurologically stable for ≥ 4 weeks).
7. Severe neurological or psychiatric disorders that might have an impact on study results in the opinion of the investigator.
8. Pregnant or lactating women or patients planning a pregnancy during the study period.
9. Participation in another clinical trial within 30 days prior to the 1st treatment.
10. History of bleeding or digestive disorders:

    * Evidence of active bleeding, bleeding diathesis, coagulopathy, or tumor with macrovascular invasion
    * Clinically significant digestive ulcer, gastrointestinal (GI) bleeding, GI or non-GI fistula, perforation, intra-abdominal abscess, clinical symptoms and signs of GI obstruction, patients requiring parenteral fluids or nutrition, history of digestive disorders such as inflammatory bowel disease
    * Evidence of pneumoperitoneum unexplained by recent surgery or paracentesis
11. Treatment with biguanides (e.g., metformin) within 2 weeks prior to the 1st treatment or anticipated required treatment with biguanides during the study period.
12. Patients requiring continuous treatment with systemic corticosteroids. However, the following will be permitted:

    - Use of local corticosteroids such as local intra-articular, intra-nasal, intra-ocular, or inhaled corticosteroids or temporary use of systemic corticosteroids for the treatment and prevention of adverse events (AEs) or allergic reactions to contrast agents will be permitted.
13. Patients with HIV and other severe diseases that would limit a patient's participation in the study in the opinion of the investigator (medically controlled diseases will be permitted).
14. Having ascites and/or pleural fluid drained within 14 days prior to screening.
15. Hemoptysis within 14 days prior to screening (≥ 1/2 teaspoonful cherry red blood per episode).
16. Core biopsy or any other minor surgical procedure within 14 days prior to initial IP dose (except for placing a vascular access).
17. Serious, unhealed scars, active ulcers, or untreated fractures.
18. History of cerebrovascular accident (stroke), transient ischemic attack, or subarachnoid hemorrhage within 6 months prior to screening.
19. History of glucose-6-phosphate dehydrogenase deficiency.
20. Individuals ineligible for this study for other reasons in the opinion of the investigator.
21. Patients identified with hypercalcemia (corrected calcium concentration > 10.4 mg/dL (2.6mmol/L)) identified during the screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose(MTD) | 4weeks
  MTD will be defined as the maximum dose level at which no more than 1 of 3 participants experience a dose-limiting toxicity (DLT) within the first 4 weeks of dosing

SECONDARY OUTCOMES:
Objective response rate(ORR) | From first dose until documented disease progression or death, up to 36 months or until database cutoff date of 14Jul2023]
  The proportion of patients achieving a partial response (PR) or complete response (CR) per RECIST 1.1
Progression Free Survival(PFS) | From first dose until documented disease progression or death, up to 36 months or until database cutoff date of 14Jul2023]
  Time from first dose until disease progression or death using RECIST 1.1
Duration of Response(DoR) | From first dose until documented disease progression or death, up to 36 months or until database cutoff date of 14Jul2023]
  Time from first PR or CR until disease progression or death using RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (2):
- California Research Institute, Los Angeles, California, United States
- Seoul national university bundang hospital, Seongnam-si, Gyeonggi-do, South Korea